CLINICAL TRIAL: NCT03344055
Title: Endocuff-assisted Colonoscopy vs Standard Colonoscopy on Adenoma Detection Rate: A Comparative Prospective Study in Common Practice
Brief Title: Endocuff-assisted Colonoscopy vs Standard Colonoscopy on Adenoma Detection Rate
Acronym: Cuff-Bercy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, KARSENTI, MD, Principal Investigator, Société Française d'Endoscopie Digestive
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A00549-44
Record Dates: First submitted 2017-11-12; First posted 2017-11-17 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Colonic Adenoma; Colonic Polyp; Colonoscopy
Keywords: Adenoma Detection Rate; Endocuff; Colonoscopy
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colonoscopy with Endocuff Vision (ECV) (Active Comparator): ECV-assisted colonoscopy ( with the use of Endocuff Vision (ECV) Second generation)
  Interventions: Device: Endocuff Vision (ECV) second generation
- Standard colonoscopy (No Intervention): Standard colonoscopy (without the use of Endocuff Vision (ECV) Second generation)

INTERVENTIONS:
Device: Endocuff Vision (ECV) second generation — Colonoscopy performed with the use of "Endocuff Vision (ECV) second generation" at the tip of the scope
  Arms: Colonoscopy with Endocuff Vision (ECV)

SUMMARY:
This is a prospective study comparing endocuff-assisted colonoscopy to standard colonoscopy. The goal of this study is to evaluate the interest of second-generation Endocuff Vision (ECV) to improve Adenoma detection rate and / or Polyp detection rate as the Mean Number of Polyps (average number of polyps) in routine colonoscopy.

This is a prospective comparative study, on 2000 patients, 1000 in each group (with and without ECV)

DETAILED DESCRIPTION:
This is a prospective study comparing endocuff-assisted colonoscopy to standard colonoscopy. The goal of this study is to evaluate the interest of second-generation Endocuff Vision (ECV) to improve Adenoma detection rate and / or Polyp detection rate as the Mean Number of Polyps (average number of polyps) in routine colonoscopy.

Number of patients:

2000 patients, 1000 in each group (with and without ECV). To limit the risk of bias, the investigators will random two teams of 12 endoscopists matched in number, volume of activity and Adenoma Detection Rate (evaluated over a period of the year preceding the study).

Both periods of study will be approximately 3-4 months in length. In order to achieve a perfect balance between the two groups of patients, an inclusion tracking chart will be initiate and will be carefully controlled. Rebalancing will be done for both periods of study to obtain 500 patients per group and per period (= 2000 patients included).

Inclusion of 500 consecutive colonoscopies in each team of investigators, a "colonoscopy with ECV" team, a "colonoscopy without ECV" team then switch and inclusion of 500 new consecutive colonoscopies in each team, ie 2000 colonoscopies in total.

The selection of the team that will begin with ECV (Team A) and the team that will finish with ECV (Team B) will be chosen at random before the start of the study.

A comparison of the two colonoscopy groups with ECV vs without ECV will be made for each team (the investigator will be his own control) and then on the overall population after the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patient scheduled for total colonoscopic exploration, during the period study
2. Patient over or equal to 18 years
3. ASA 1, ASA 2, ASA 3
4. No participation in another clinical study
5. Certificate of non opposition signed

Exclusion Criteria:

1. Patient under 18 years old
2. ASA 4, ASA 5
3. Pregnant woman
4. Patient with coagulation abnormalities preventing polypectomy: prothrombin level <50%, Platelets <50000 / mm3, effective anti-coagulation in progress, clopidogrel in progress.
5. Inflammatory bowel disease
6. Known colonic stenosis
7. Diverticulitis less than 6 weeks old
8. Patient unable to give consent or protected by law
9. Opposition expressed for inclusion in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2059 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate (ADR) | during procedure
  rate (%) of colonoscopies with one or more adenoma detected

SECONDARY OUTCOMES:
Polyp detection rate (PDR) | during procedure
  rate (%) of colonoscopies with one or more polyp detected
Advanced neoplasia detection rate (ANDR) | during procedure
  rate (%) of colonoscopies with one or more advanced neoplasia detected
Serrated polyp detection rate (SPDR) | during procedure
  rate (%) of colonoscopies with one or more serrated polyp detected
Morbidity: perforation rate (%) | 21 days after procedure
  Perforation rates (%)
Morbidity: bleeding rate (%) | 21 days after procedure
  Bleeding rates (%)
caecal intubation rate (%) | during procedure
  caecal intubation rate (complete colonoscopy)
Time to reach caecum (sec) | during procedure
  Time to reach caecum from the beginning of the procedure (in seconds)
withdrawal time (sec) | during procedure
  withdrawal time of the scope from the caecum to the end of the procedure (in seconds)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique PARIS-BERCY, Charenton-le-Pont, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karsenti D, Tharsis G, Perrot B, Cattan P, Tordjman G, Venezia F, Zrihen E, Gillot D, Gillet A, Hagege C, Samama J, Etienney I, Lab JP, Guigui B, Zago J, Benkessou B, Burtin P, Cavicchi M. Adenoma detection by Endocuff-assisted versus standard colonoscopy in routine practice: a cluster-randomised crossover trial. Gut. 2020 Dec;69(12):2159-2164. doi: 10.1136/gutjnl-2019-319565. Epub 2020 Mar 24. PMID 32209605